CLINICAL TRIAL: NCT04603846
Title: A Study of Anti-PD-L1 Antibody ZKAB001 Combined With Albumin-bound Paclitaxel in Advanced Urothelial Carcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTL-LEES-2019-06
Record Dates: First submitted 2020-09-08; First posted 2020-10-27 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Advanced Urothelial Carcinoma
MeSH Terms: interventions — Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined treatment group (Experimental): All patients will receive 16 cycles of anti-PD-L1 antibody (5mg/kg, IV, every 3 weeks) , concurrently with 6 cycles of albumin-bound paclitaxel 260mg/m2 d1，q3w；
  Interventions: Drug: anti-PD-L1 antibody; Drug: albumin bound paclitaxel

INTERVENTIONS:
Drug: anti-PD-L1 antibody — Patients will receive 16 cycles of anti-PD-L1 antibody 5mg/kg IV on day 1 every 3 weeks.
  Other Names: ZKAB001
Drug: albumin bound paclitaxel — Patients will receive 6 cycles of albumin bound paclitaxel 260mg/m2 on days 1 every 3 weeks .
  Other Names: ABRAXANE

SUMMARY:
To evaluate the safety and efficacy of recombinant anti-PD-L1 monoclonal antibody injection (ZKAB001) combined with Albumin-bound paclitaxel in the treatment of Advanced urothelial carcinoma

DETAILED DESCRIPTION:
This trial is designed to first include 6 subjects to confirm the dose safety. If the toxicity is intolerable, the dose of chemotherapeutic drugs will be reduced depending on the toxicity for further exploration.If it was tolerated, the recommended dose was determined, and the dose was extended. 14 patients were enrolled to further observe the safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old;
* Pathologically confirmed urothelial carcinoma;
* Terminal patients who have not received treatment or for the first time recurrence more than 6 months after the end of adjuvant chemotherapy after surgery;
* Evaluable lesions based on RECIST V1.1;
* ECOG score 0-1;
* Estimated life expectancy >3 months;
* The function of important organs meets the following requirements;
* The subjects voluntarily joined the study, signed informed consent, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

* Previously received drugs targeting PD-1, PD-L1, PD-L2 or other treatments targeting T cell costimulation or checkpoint channels;
* Received systemic corticosteroid immunosuppressants 2 weeks before the study;
* Suffer from active meningeal metastasis or uncontrolled, untreated brain metastasis;
* Severe cardiovascular disease, such as New York Heart Association (New York Heart Association,NYHA standard) Grade 3-4 heart failure, unstable angina pectoris, unstable arrhythmia, or color heart photo indicates LVEF (left ventricular ejection fraction) < 50%;
* Previous hypersensitivity to monoclonal antibodies;
* The patient has known, active or suspected autoimmune diseases. The following conditions are allowed: skin diseases that do not require systemic treatment (such as vitiligo, psoriasis), type I diabetes, autoimmune hypothyroidism with hormone replacement therapy;
* The study drug suffered from other active malignant tumors within 5 years before the first use of the drug. Cured localized tumors, such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the prostate, carcinoma in situ of the cervix, carcinoma in situ of the breast, etc., can be included in the group;
* Active hepatitis B or C (unless HBV-DNA titer < 500IU/mL or copy number < 1000copies/ml, HCV-RNA negative after antiviral treatment can be included in), HIV positive or known history of acquired immunodeficiency syndrome;
* Severe infection existed before screening, including but not limited to, infections requiring hospitalization, bacteremia, severe pneumonia, etc;
* There has been active pulmonary tuberculosis in the past year, whether treated or not;
* Live attenuated vaccine was used within 28 days prior to screening;
* Patients who have previously received allogeneic bone marrow transplantation or solid organ transplantation;
* Have received any other experimental drug treatment within 28 days prior to signing ICF;
* Pregnant or lactating women;
* Patients of childbearing age who refuse to use effective contraception;
* Other researchers believe that it is not suitable to join the group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-08-25 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 21 days after first dose
  Adverse events of level 3 or above related to the study drug occurring within 21 days after the first dose as assessed by CTCAE v5.0.
Recommended phase II dose (RP2D) | 21 days after first dose
  DLT occurs in no more than 1/6 subjects, this dose is defined as RP2D.

SECONDARY OUTCOMES:
objective response rate | 12 months
  Percentage of patients in partial and complete response
progression free survival | 12 months
  time between first dose of study drug to disease progression
PD-L1 expression | 12 months
  The positive rate of PD-L1 expression in tumor tissue.
TMB expression | 12 months
  The positive rate of TMB expression in tumor tissue.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tumor Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tang B, Xiao J, Chi Z, Duan R, Cui C, Si L, Liu Y, Hu X, Liu Z, Xiang P, Li S, Yan X, Zhou L, Li J, Li Y, Yu X, Dai X, Li X, Guo J, Sheng X. Phase Ib study of anti-PD-L1 monoclonal antibody socazolimab in combination with nab-paclitaxel as first-line therapy for advanced urothelial carcinoma. Oncologist. 2025 Feb 6;30(2):oyae260. doi: 10.1093/oncolo/oyae260. PMID 39418340